CLINICAL TRIAL: NCT02424500
Title: Prospective, Open-Label, Randomized, Controlled, Multi-Center Study Comparing Efficacy and Safety of Frequently Modified Insulin Therapy Using Dosage Recommending Device
Brief Title: Multi-Center Study Comparing Efficacy and Safety of Frequently Modified Insulin Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hygieia Research LLC (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PD004-1; 5R42DK085974-03 (NIH)
Record Dates: First submitted 2015-04-09; First posted 2015-04-23 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus, Type 2; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- d-Nav Device (Experimental): d-Nav Device: daily use to provide insulin dosage updates weekly - or sooner when needed based on analyzes and evaluates the historical blood glucose patterns.
  Insulin dosage is adjusted as required
  Interventions: Device: d-Nav
- Blood Glucose Monitoring System (Active Comparator): Patient's personal Over the Counter Blood Glucose Monitoring System (OTC BGMS) for daily glucose testing to determine insulin dosage needed.
  Insulin dosage is adjusted as required
  Interventions: Device: Blood Glucose Monitoring System

INTERVENTIONS:
Device: d-Nav — Insulin dosage is adjusted as required
  Arms: d-Nav Device
Device: Blood Glucose Monitoring System — Insulin dosage is adjusted as required
  Arms: Blood Glucose Monitoring System

SUMMARY:
Hygieia Research seeks to conduct a prospective randomized clinical study involving adult subjects with uncontrolled Type-2 diabetes requiring insulin. The study seeks to demonstrate that the clinical application of the d-Nav will achieve metabolic control in a safe and effective manner.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate that the use of d-Nav (d-Nav group) is superior to titration of insulin dosage relying on data from glucose meters with health care provider support (Control) in the management of insulin treated diabetes, by randomizing 200 insulin treated subjects with type 2 diabetes.

Primary Objective: To demonstrate a greater reduction in HbA1c at 6-months for d-Nav users compared to control patients in the primary cohort.

ELIGIBILITY:
Inclusion Criteria:

1. 21 to 70 years of age
2. If female, must be of non-childbearing potential or have a negative urine pregnancy test at screening and using adequate method of contraception throughout conduct of the study
3. Clinical diagnosis of Type-2 diabetes for at least 1-year
4. HbA1c 7.5% to 11% inclusive
5. Total daily dose of insulin of 25 units or more (10 units if on Lantus® alone) using one of these insulin regimens:

   * Regimen 1 - a single injection of the long-acting insulin analog Lantus® (Glargine) per day (limited to a daily dose that is no more than 0.7 units per kg of body weight);
   * Regimen 2 - twice daily biphasic insulin (i.e., Humalog® Mix 75/25, NovoLog® Mix 70/30) or pre-mixed insulin (i.e., Humulin® 70/30, Novolin® 70/30);
   * Regimen 3 - a short-acting insulin analog (i.e., Humalog®-Lispro, NovoLog®-Aspart, Apidra®-Glulisine) before each meal and are treated with a single injection of the long-acting insulin analog Lantus® (Glargine) per day and do not utilize an insulin/carbohydrate ratio for calculating their short-acting insulin doses; or
   * Regimen 4 - with a short-acting insulin analog (i.e., Humalog®-Lispro, NovoLog®-Aspart, Apidra®-Glulisine) before each meal and a single injection of the long-acting insulin analog Lantus® (Glargine) per day and utilize an insulin/carbohydrate ratio for calculating their short-acting insulin doses.
6. On same insulin regimen for the previous 3-months
7. May be using other diabetes agents at a stable dose for the last 3-months
8. Signed and dated informed consent document, which contains HIPAA waiver information informing about all of the aspects of the clinical study;
9. Will regularly conduct Self-Monitored Blood Glucose. Prior to randomization must meet the following .

   Minimum number of tests required from all subjects:
   * Basal insulin subjects at least 4 fasting glucose readings/wk
   * Premixed insulin subjects at least 8 readings/wk
   * Basal-bolus insulin therapy subjects at least 16 total readings/wk
10. Willing and able to comply with the scheduled clinical study activities and glucose testing:

    * Basal insulin subjects at least 5 fasting glucose readings/wk
    * Premixed insulin subjects at least 5 pre-breakfast and 5 pre-evening meal readings/wk
    * Basal-bolus insulin therapy subjects at least 20 total readings/wk which include 5 readings before each of the following time points: breakfast, lunch, evening meal and bedtime.

    Note: All subjects may be asked to test during the night if clinically indicated.
11. Participant must have a primary care provider

Exclusion Criteria:

1. History >2 episodes of severe hypoglycemia (see definition below) in the past year, or hypoglycemic unawareness when glucose levels are ≤ 50 mg/dl;
2. Significant physical, psychological, or cognitive impairment that would prohibit adherence to the protocol at the discretion of the PI;
3. Splitting Lantus and taking Lantus twice a day
4. Severe cardiovascular disease including a history of congestive heart failure, unstable angina, myocardial infarction or stroke within the 6-months preceding enrollment;
5. Active anemia w/ hematocrit ≤ 25% in women or 30% in men;
6. Advanced kidney disease Stage 4 (eGFR < 30 ml/min) and above
7. Active cancer or cancer in the past 2-years (except non-melanoma skin cancer)
8. History of significant liver disease including cirrhosis or elevated liver enzymes (e.g., AST and ALT greater than 3 times the upper limit of normal values).
9. BMI > 45 kg/m2
10. Are pregnant, plan to become pregnant during the study period, or are breastfeeding.
11. Have a BGMS that cannot be downloaded.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2015-01; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Reduction in HbA1C | 6 months
  To demonstrate a greater reduction in HbA1c at 6-months for d-Nav users compared to control patients in the primary cohort.

SECONDARY OUTCOMES:
Comparison Percent Reduction HbA1c | 6 months
  To determine the difference between the Control and d-Nav group in the percent of participants who achieve A1c < 7.0%, < 8.0%, and >9.0% at 6 months
Number of Glucose Readings <70 mg/dl | 3 and 6 months
  To determine the difference between the Control and d-Nav group in the number of glucose readings <70 mg/dl (symptomatic or asymptomatic) utilizing the documented downloaded glucose values.
Change in Rate of Hypoglycemia | 6 months
  To determine change (if any) in rate of hypoglycemia, during the study for d-Nav users in the secondary cohort
Comparison Percent Reduction HbA1c w/out Hypoglycemia | 6 months
  To determine the difference between the Control and d-Nav group in the percent of participants who achieve A1c < 7.0%, < 8.0% without a severe hypoglycemia event at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Bergenstal, MD, Principal Investigator — Executive Director International Diabetes Center
Locations (1):
- Park Nicollet Institute / International Diabetes Center, Minneapolis, MN, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Bergenstal RM, Johnson M, Passi R, Bhargava A, Young N, Kruger DF, Bashan E, Bisgaier SG, Isaman DJM, Hodish I. Automated insulin dosing guidance to optimise insulin management in patients with type 2 diabetes: a multicentre, randomised controlled trial. Lancet. 2019 Mar 16;393(10176):1138-1148. doi: 10.1016/S0140-6736(19)30368-X. Epub 2019 Feb 23. PMID 30808512